CLINICAL TRIAL: NCT00983866
Title: Increasing Participation in Cancer Clinical Trials
Brief Title: CHOICES: Understanding Clinical Trials as a Treatment Option
Acronym: CHOICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CN-04CSomk-02-B; R01CA114543 (NIH)
Record Dates: First submitted 2009-09-14; First posted 2009-09-24 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored Telephone Counseling (Experimental)
  Interventions: Behavioral: Tailored Telephone Counseling
- Standard Trial Recruitment Procedures (No Intervention)

INTERVENTIONS:
Behavioral: Tailored Telephone Counseling — The intervention is comprised of a letter introducing patients to the idea of participating in a clinical trial as a possible treatment option, followed by a telephone call by a nurse educator who describes the clinical trials process and answers any questions patients may have. The nurse educators will use a tailored counseling protocol that will enable them to conduct an assessment of patients' understanding about and interest in clinical trials and tailor messages according to patient health literacy and language. The protocol will consist of both proactive and reactive counseling. The nurse educator will have a general list of topics to cover but will tailor the discussion and information provided to individual patients' questions and desire for particular types of information.
  Arms: Tailored Telephone Counseling

SUMMARY:
The goal of this study is to determine whether having a telephone discussion with a nurse educator about making treatment decisions and participating in a clinical trial increases trial participation.

The investigators hypothesize that the participants in the intervention group will be more likely to take part in a clinical trial than those in the usual care group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are potentially eligible for one of the designated clinical trials on the basis of automated data from pathology reports and other databases

Exclusion Criteria:

* Patients who meet specific exclusion criteria for designated clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1376 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients eligible for designated clinical trials who actually enroll in one of these trials | Up to three months after the index oncology visit

SECONDARY OUTCOMES:
Proportion of patients who leave the identification and recruitment process at each step. | Up to three months after the index oncology visit

CONTACTS AND LOCATIONS:
Overall Officials: Lou Fehrenbacher, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States